CLINICAL TRIAL: NCT01372410
Title: A Randomized, Double Blind, Placebo Controlled, Incomplete Block, Crossover, Dose Ranging Study to Evaluate the Dose Response of GSK573719 Administered Once or Twice Daily Over 7 Days in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: AC4115321
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 115321
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Long acting muscarinic antagonist; Tiotropium; Chronic Bronchitis; Emphysema; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — GSK573719; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tiotropium (Active Comparator): 18 mcg, inhaled long acting muscarinic antagonist
  Interventions: Drug: Tiotropium
- GSK573719 (Experimental): inhaled medication
  Interventions: Drug: GSK573719
- Placebo (Placebo Comparator): inactive/excipients only
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK573719 — 125 mcg once daily
  Arms: GSK573719
Drug: GSK573719 — 62.5 mcg once daily
  Arms: GSK573719
Drug: GSK573719 — 31.25 mcg once daily
  Arms: GSK573719
Drug: GSK573719 — 15.6 mcg once daily
  Arms: GSK573719
Drug: GSK573719 — 31.25 mcg twice daily
  Arms: GSK573719
Drug: GSK573719 — 15.6 mcg twice daily
  Arms: GSK573719
Drug: Tiotropium — 18 mcg once daily
  Arms: Tiotropium
Drug: Placebo — once or twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to further characterize the dose response of GSK573719 at doses of 15.6 micrograms (mcg) to 125 mcg once daily in patients with chronic obstructive pulmonary disease (COPD). Treatment with doses of GSK573719 dosed twice daily will also be included to further evaluate dosing frequency. Treatment with tiotropium (18 mcg) once daily via the Handihaler will be included as an active control. A placebo treatment will be included in order to evaluate absolute treatment effect of the different doses of GSK573719.

DETAILED DESCRIPTION:
Inhaled bronchodilators, such as beta 2 agonists and anticholinergics, and inhaled corticosteroids are the mainstays of therapy in patients diagnosed with COPD. Anticholinergic bronchodilators or long acting muscarinic receptor antagonists function by blocking endogenous airway smooth muscle cholinergic tone. Treatment with anticholinergics has been shown to significantly improve forced expiratory volume in 1 second (FEV1), resting and dynamic lung hyperinflation, symptoms, and exercise capacity in patients with COPD. Currently tiotropium is the only approved long acting muscarinic antagonist available for treatment of COPD.

This is a multicenter, randomized, double-blind, placebo controlled, three way crossover, incomplete block study to evaluate 4 doses of GSK573719 inhaled once daily and 2 doses of GSK573719 inhaled twice daily over 7 days in patients with COPD. Tiotropium will be included as an open label active comparator. A placebo treatment will be included to evaluate treatment effect of each GSK573719 dose. Pharmacokinetic profiles of GSK573719 will also be determined. Each eligible subject will receive a sequence of 3 of 8 potential treatments for a total of 3 treatment periods per subject. There will be 7 clinic visits, during three of which 24 hour serial spirometry will be performed. The total duration of subject participation is approximately 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient
* A signed and dated written informed consent prior to study participation.
* Male or female adults.
* 40 to 80 years of age at Visit 1
* Diagnosis of COPD
* Current or former cigarette smokers with a history of cigarette smoking of greater than or equal to 10 pack-years
* Post-albuterol forced expiratory volume in 1 second (FEV1)/ forced vital capacity (FVC)<0.70 and post albuterol FEV1 of greater than or equal to 35% and less than or equal to 70% of predicted normal values

Exclusion Criteria:

* Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* A current diagnosis of asthma
* Known alpha-1 antitrypsin deficiency, active lung infections (such as tuberculosis), and lung cancer
* Other significant respiratory conditions in addition to COPD
* Other diseases that are uncontrolled including cancer in remission for less than 5 years
* Chest x-ray or CT scan with clinically significant abnormalities not believed to be due to the presence of COPD
* Hypersensitivity to any anticholinergic/muscarinic receptor antagonist, beta2-agonist, lactose/milk protein or magnesium stearate
* A medical condition that contraindicates study participation or use of an inhaled anticholinergic
* Hospitalization for COPD or pneumonia within 12 weeks of Visit 1
* Any previous lung resection surgery
* A body mass index (BMI) value of >35 kilogram (kg)/meter squared (m2)
* An abnormal and significant electrocardiogram finding at Visit 1
* Significantly abnormal finding from clinical chemistry or haematology tests at Visit 1.
* A positive Hepatitis B surface antigen or positive Hepatitis C antibody
* Medically unable to withhold albuterol (salbutamol) for the 6 hour period prior to study visits
* Use of depot corticosteroids within 12 weeks of Visit 1
* Use of oral or parenteral corticosteroids or antibiotics for lower respiratory tract infection within 6 weeks of Visit 1
* Use of long-acting beta-agonist (LABA)/inhaled corticosteroid (ICS) product if LABA/ICS therapy is discontinued within 30 days of Visit 1
* Use of ICS at a dose of >1000mcg/day of fluticasone propionate or equivalent within 30 days of Visit 1
* Initiation or discontinuation of ICS within 30 days of Visit 1
* Use of tiotropium or phosphodiesterase 4 inhibitors within 14 days of Visit 1
* Use of theophyllines, oral leukotriene inhibitors, long-acting oral beta-agonists, or inhaled long-acting beta-agonists within 48 hours of Visit 1
* Short-acting oral beta-agonists within 12 hours of Visit 1
* Use of LABA/ICS combination products only if discontinuing LABA therapy and switching to ICS monotherapy within 48 hours of Visit 1 for the LABA component
* Use of sodium cromoglycate or nedocromil sodium within 24 hours of Visit 1
* Use of inhaled short-acting beta-agonists, inhaled short-acting anticholinergics, or inhaled short-acting anticholinergic/short-acting beta-agonist combination products within 6 hours of Visit 1
* Use of any other investigational medication within 30 days or 5 drug half-lives (whichever is longer)
* Oxygen therapy prescribed for greater than 12 hours a day
* Regular use (prescribed for use every day, not for as-needed use) of short-acting bronchodilators
* Use of continuous positive airway pressure (CPAP), nocturnal positive pressure or non-invasive positive pressure ventilation (NIPPV), including use for sleep apnea.
* Acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1
* A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1
* Anyone affiliated with investigator site
* Previous use of GSK573719 or GSK53719/GW642444

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2011-07-01; Primary Completion 2011-10-01 (Actual); Study Completion 2011-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- United States (13):
  - GSK Investigational Site, Costa Mesa, California
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Duluth, Georgia
  - GSK Investigational Site, Edina, Minnesota
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Church A, Beerahee M, Brooks J, Mehta R, Shah P. Dose response of umeclidinium administered once or twice daily in patients with COPD: a randomised cross-over study. BMC Pulm Med. 2014 Jan 6;14:2. doi: 10.1186/1471-2466-14-2. PMID 24393134
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 115321 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115321 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115321 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115321 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115321 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115321 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115321 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to receive a sequence of 3 of 8 possible treatments over 3 treatment periods. There are 56 combinations of 3 treatments from the 8 study treatments, each of which can be ordered in 6 ways (totaling 336 possible sequences; 163 were randomly assigned). Participant Flow data are presented by treatment rather than sequence.
Groups:
- Placebo: Participants received matching placebo once in the morning and once in the evening for 7 days via a dry powder inhaler (DPI) in one of three 7-day treatment periods. Treatment Periods 1 and 2 were followed by a 10- to 14-day Washout Period; Treatment Period 3 was followed by a 7- to 9-day Washout Period before the follow-up phone call.
- UMEC 15.6 µg QD: Participants received an inhaled dose of a dry powder formulation of umeclidinium bromide (UMEC) 15.6 micrograms (µg) once a day (QD) for 7 days in the morning, and matching placebo QD for 7 days in the evening, via a DPI in one of three 7-day treatment periods. Treatment Periods 1 and 2 were followed by a 10- to 14-day Washout Period; Treatment Period 3 was followed by a 7- to 9-day Washout Period before the follow-up phone call.
- UMEC 31.25 µg QD: Participants received an inhaled dose of a dry powder formulation of UMEC 31.25 µg QD for 7 days in the morning, and matching placebo QD for 7 days in the evening, via a DPI in one of three 7-day treatment periods. Treatment Periods 1 and 2 were followed by a 10- to 14-day Washout Period; Treatment Period 3 was followed by a 7- to 9-day Washout Period before the follow-up phone call.
- UMEC 62.5 µg QD: Participants received an inhaled dose of a dry powder formulation of UMEC 62.5 µg QD for 7 days in the morning, and matching placebo QD for 7 days in the evening, via a DPI in one of three 7-day treatment periods. Treatment Periods 1 and 2 were followed by a 10- to 14-day Washout Period; Treatment Period 3 was followed by a 7- to 9-day Washout Period before the follow-up phone call.
- UMEC 125 µg QD: Participants received an inhaled dose of a dry powder formulation of UMEC 125 µg QD for 7 days in the morning, and matching placebo QD for 7 days in the evening, via a DPI in one of three 7-day treatment periods. Treatment Periods 1 and 2 were followed by a 10- to 14-day Washout Period; Treatment Period 3 was followed by a 7- to 9-day Washout Period before the follow-up phone call.
- UMEC 15.6 µg BID: Participants received an inhaled dose of a dry powder formulation of UMEC 15.6 µg once in the morning and once in the evening for 7 days via a DPI in one of three 7-day treatment periods. Treatment Periods 1 and 2 were followed by a 10- to 14-day Washout Period; Treatment Period 3 was followed by a 7- to 9-day Washout Period before the follow-up phone call.
- UMEC 31.25 µg BID: Participants received an inhaled dose of a dry powder formulation of UMEC 31.25 µg once in the morning and once in the evening for 7 days via a DPI in one of three 7-day treatment periods. Treatment Periods 1 and 2 were followed by a 10- to 14-day Washout Period; Treatment Period 3 was followed by a 7- to 9-day Washout Period before the follow-up phone call.
- TIO 18 µg QD: Participants received tiotropium bromide (TIO) 18 µg inhalation capsules via the HandiHaler dry powder inhaler for 7 days in the morning and placebo via the DPI in the evening in one of three 7-day treatment periods. Treatment Periods 1 and 2 were followed by a 10- to 14-day Washout Period; Treatment Period 3 was followed by a 7- to 9-day Washout Period before the follow-up phone call.
Period: Treatment Period 1 (7 Days)
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID | TIO 18 µg QD
Started | 20 | 21 | 19 | 20 | 21 | 21 | 22 | 19
Completed | 19 | 19 | 19 | 20 | 19 | 21 | 20 | 19
Not Completed | 1 | 2 | 0 | 0 | 2 | 0 | 2 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Participant Withdrew Consent | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Washout Period 1 (10-14 Days)
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID | TIO 18 µg QD
Started | 19 | 19 | 19 | 20 | 19 | 21 | 20 | 19
Completed | 18 (Participants withdrawing during washout are counted under the last treatment taken.) | 19 (Participants withdrawing during washout are counted under the last treatment taken.) | 19 (Participants withdrawing during washout are counted under the last treatment taken.) | 20 (Participants withdrawing during washout are counted under the last treatment taken.) | 19 (Participants withdrawing during washout are counted under the last treatment taken.) | 21 (Participants withdrawing during washout are counted under the last treatment taken.) | 20 (Participants withdrawing during washout are counted under the last treatment taken.) | 18 (Participants withdrawing during washout are counted under the last treatment taken.)
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Participant Withdrew Consent | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment Period 2 (7 Days)
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID | TIO 18 µg QD
Started | 19 (By crossover design, participants were assigned to a different treatment arm in each period.) | 21 (By crossover design, participants were assigned to a different treatment arm in each period.) | 22 (By crossover design, participants were assigned to a different treatment arm in each period.) | 17 (By crossover design, participants were assigned to a different treatment arm in each period.) | 19 (By crossover design, participants were assigned to a different treatment arm in each period.) | 16 (By crossover design, participants were assigned to a different treatment arm in each period.) | 21 (By crossover design, participants were assigned to a different treatment arm in each period.) | 19 (By crossover design, participants were assigned to a different treatment arm in each period.)
Completed | 19 | 21 | 22 | 17 | 19 | 16 | 21 | 19
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (10-14 Days)
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID | TIO 18 µg QD
Started | 19 | 21 | 22 | 17 | 19 | 16 | 21 | 19
Completed | 19 (Participants withdrawing during washout are counted under the last treatment taken.) | 21 (Participants withdrawing during washout are counted under the last treatment taken.) | 22 (Participants withdrawing during washout are counted under the last treatment taken.) | 17 (Participants withdrawing during washout are counted under the last treatment taken.) | 17 (Participants withdrawing during washout are counted under the last treatment taken.) | 16 (Participants withdrawing during washout are counted under the last treatment taken.) | 20 (Participants withdrawing during washout are counted under the last treatment taken.) | 17 (Participants withdrawing during washout are counted under the last treatment taken.)
Not Completed | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Participant Withdrew Consent | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment Period 3 (7 Days)
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID | TIO 18 µg QD
Started | 21 (By crossover design, participants were assigned to a different treatment arm in each period.) | 18 (By crossover design, participants were assigned to a different treatment arm in each period.) | 16 (By crossover design, participants were assigned to a different treatment arm in each period.) | 22 (By crossover design, participants were assigned to a different treatment arm in each period.) | 20 (By crossover design, participants were assigned to a different treatment arm in each period.) | 19 (By crossover design, participants were assigned to a different treatment arm in each period.) | 15 (By crossover design, participants were assigned to a different treatment arm in each period.) | 18 (By crossover design, participants were assigned to a different treatment arm in each period.)
Completed | 21 | 18 | 15 | 22 | 20 | 18 | 15 | 18
Not Completed | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Treatments: Participants received a sequence containing 3 of the following 8 possible treatments: placebo; UMEC 15.6 µg, 31.25 µg, 62.5 µg, and 125 µg QD; UMEC 15.6 µg and 31.25 µg BID; TIO 18 µg QD. Participants received each of the treatments in 1 of 3 7-day treatment periods, each of which was followed by a Washout Period. Treatment Periods 1 and 2 were followed by a 10- to 14-day Washout Period; Treatment Period 3 was followed by a 7- to 9-day Washout Period before the follow-up phone call.
Arm/Group | All Study Treatments
Number analyzed (Participants) | 163
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.5 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 78
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 16
  American Indian or Alaska Native | 1
  White - White/Caucasian/European Heritage | 145
  Mixed Race | 1

OUTCOME MEASURES:

1. Primary Outcome: Final Dose-response Model for Trough Forced Expiratory Volume in One Second (FEV1)
Description: The trough FEV1 data for both the once-daily (QD) and twice-daily (BID) UMEC doses were included in a parametric analysis in order to evaluate trough FEV1dose response. The Day 8 dataset and a pooled dataset for Day 7 and Day 8 were analyzed separately and reported. The rationale for pooling Day 7 and Day 8 (post-hoc analysis) was to ensure informative interpretation of FEV1 response as a function of dose given the repeated measures for trough FEV1 response within each participant on different days. The fixed-effects parameters of the dose response model include Emax (the maximum predicted FEV1 response), ED50 (potency), and S0 (estimated Baseline FEV1). FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Data for Emax and S0 are reported in this table. mITT=Modified Intent-to-Treat; par.=participants; BL=Baseline.
Time Frame: Day 7 and Day 8 of each treatment period (up to Study Day 50)
Population: mITT Population: par. randomized to treatment who received >=1 dose of study medication. Par. with >=1 post-BL assessment and non-missing covariate data are included in the analysis. Different par. may have been analyzed at different time points (n=X in category titles); the overall number of par. analyzed reflects everyone in the mITT Population.
Measure: Geometric Mean (95% Confidence Interval); unit: Liters
Arm/Group | All Study Treatments
Number analyzed (Participants) | 163
Liters
  Day 8, Emax, n=157 | 0.185 [0.154 to 0.216]
  Pooled Day 7 and Day 8, Emax, n=160 | 0.156 [0.123 to 0.189]
  Day 8, S0, n=157 | 1.24 [1.21 to 1.27]
  Pooled Day 7 and 8, S0, n=160 | 1.24 [1.21 to 1.27]

2. Secondary Outcome: Change From Baseline (BL) in Serial FEV1 Over Time on Day 7 of Each Treatment Period
Description: Serial FEV1 for once daily dosing is recorded at the pre-AM dose (AMD; time 0 hour [h]) and at 1, 3, 6, 9, 12,13, 15, 23, and 24 hours after the AMD on Day 7. For twice daily dosing, the 12 h AMD corresponds to the pre-PM dose (PMD), the 13 h AMD corresponds to the 1 h PMD, the 15 h AMD corresponds to the 3 h PMD, the 23 h AMD corresponds to the 11 h PMD, and the 24 h AMD corresponds to the 12 h PMD in this table. Analysis was performed using a mixed model with covariates of mean BL, period BL, treatment, period, time, time by period BL interaction, time by mean BL interaction, and time by treatment interaction as fixed effects and participant as a random effect. BL is the value recorded pre-dose on Day 1 of each TP, mean BLis the mean of the BLs for each participant, and period BL is the difference between the BL and the mean BL in each TP for each participant. Change from BL for each timepoint within a TP is the serial FEV1 measure at that timepoint minus the BL value for that TP.
Time Frame: Baseline and Day 7 of each treatment period (TP; up to Study Day 49)
Population: mITT Population. All participants (par.) with >=1 post-BL assessment and non-missing covariate data are included in the analysis. Different par. may have been analyzed at different time points (n=X, X, X, X in the category titles), so the overall number of par. analyzed reflects everyone in the mITT Population with data available at >=1 time point.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID | TIO 18 µg QD
Number analyzed (Participants) | 60 | 59 | 56 | 59 | 60 | 55 | 57 | 56
Liters
  Pre-AMD, n=59, 58, 55, 59, 60, 54, 57, 54 | -0.007 (0.021) | 0.068 (0.021) | 0.067 (0.021) | 0.065 (0.021) | 0.122 (0.021) | 0.069 (0.022) | 0.097 (0.021) | 0.084 (0.022)
  1 h AMD, n=59, 59, 56, 59, 60, 55, 57, 56 | -0.006 (0.023) | 0.086 (0.023) | 0.112 (0.023) | 0.107 (0.023) | 0.167 (0.023) | 0.128 (0.024) | 0.135 (0.023) | 0.176 (0.023)
  3 h AMD, n=59, 59, 56, 59, 59, 55, 57, 56 | -0.013 (0.024) | 0.082 (0.024) | 0.132 (0.024) | 0.082 (0.024) | 0.176 (0.024) | 0.126 (0.025) | 0.120 (0.024) | 0.180 (0.025)
  6 h AMD, n=59, 59, 55, 59, 59, 55, 57, 56 | -0.054 (0.022) | 0.056 (0.022) | 0.067 (0.022) | 0.056 (0.022) | 0.088 (0.022) | 0.045 (0.022) | 0.081 (0.022) | 0.128 (0.022)
  9 h AMD, n=59, 59, 56, 59, 58, 55, 56, 56 | -0.072 (0.022) | 0.040 (0.022) | 0.050 (0.022) | 0.084 (0.022) | 0.132 (0.022) | 0.070 (0.023) | 0.038 (0.022) | 0.094 (0.023)
  12 h AMD/Pre-PMD, n=59, 59, 56, 59, 59, 55, 57, 56 | -0.086 (0.023) | 0.022 (0.023) | 0.028 (0.023) | 0.043 (0.023) | 0.103 (0.023) | 0.048 (0.023) | 0.048 (0.023) | 0.081 (0.023)
  13 h AMD/1 h PMD, n=59, 59, 56, 59, 58, 55, 57, 56 | -0.085 (0.024) | -0.001 (0.024) | -0.003 (0.024) | 0.026 (0.024) | 0.103 (0.024) | 0.063 (0.025) | 0.041 (0.024) | 0.061 (0.025)
  15 h AMD/3 h PMD, n=59, 58, 56, 58, 59, 55, 57, 56 | -0.112 (0.023) | -0.008 (0.023) | 0.004 (0.023) | 0.022 (0.023) | 0.073 (0.023) | 0.041 (0.024) | 0.047 (0.023) | 0.037 (0.023)
  23 h AMD/11 h PMD, n=59, 57, 56, 59, 59, 55, 57,56 | -0.101 (0.024) | 0.006 (0.025) | -0.006 (0.025) | 0.012 (0.024) | 0.073 (0.024) | 0.001 (0.025) | 0.33 (0.025) | 0.002 (0.025)
  24 h AMD/12 h PMD, n=59, 58, 56, 59, 59, 55, 57,56 | -0.065 (0.024) | 0.070 (0.024) | 0.065 (0.024) | 0.067 (0.023) | 0.146 (0.024) | 0.083 (0.024) | 0.084 (0.024) | 0.049 (0.024)

3. Secondary Outcome: Change From Baseline (BL) in Weighted Mean FEV1 Over 0 to 24 Hours After the Morning Dosing on Day 7 of Each Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. The weighted mean FEV1 was derived by calculating the area under the FEV1/time curve (AUC) using the trapezoidal rule, and then dividing the value by the time interval over which the AUC was calculated. The weighted mean FEV1 was calculated using 0-24 hour post-dose measurements at Day 7 of each treatment period, which included pre-dose and post-dose 1, 3, 6, 9, 12, 13, 15, 23, and 24 hours. Analysis was performed using a mixed model with covariates of mean BL, period BL, treatment, and period as fixed effects and participant as a random effect. BL is the FEV1 value recorded pre-dose on Day 1 of each TP, mean BL is the mean of the BLs for each participant, and period BL is the difference between the BL and the mean BL in each TP for each participant. Change from BL for each TP is the weighted mean FEV1 at Day 7 minus the BL value for that TP.
Time Frame: Baseline and Day 7 of each treatment period (TP; up to Study Day 49)
Population: mITT Population. All participants with >=1 post-Baseline assessment and non-missing covariate data are included in the analysis. The number of participants represents participants who provided data at Day 7.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID | TIO 18 µg QD
Number analyzed (Participants) | 54 | 56 | 51 | 54 | 56 | 52 | 55 | 53
Liters | -0.074 (0.018) | 0.043 (0.018) | 0.045 (0.019) | 0.059 (0.018) | 0.100 (0.018) | 0.062 (0.018) | 0.068 (0.018) | 0.084 (0.018)

4. Primary Outcome: Final Dose-response Model for Trough FEV1 for ED50 (Potency) Parameter
Description: The trough FEV1 data for both the once-daily (QD) and twice-daily (BID) UMEC doses were included in a parametric analysis in order to evaluate dose response. Both a Day 8 dataset and a pooled dataset for Day 7 and Day 8 were analyzed and reported. The rationale for pooling Day 7 and Day 8 (post-hoc analysis) was to ensure informative interpretation of FEV1 response as a function of dose given the repeated measures for trough FEV1 response within each participant on different days. ED50 is defined as the potency and is the dose that yields 50% of Emax (maximum predicted FEV1 response). FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second.
Time Frame: Day 7 and Day 8 of each treatment period (up to Study Day 50)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms
Arm/Group | All Study Treatments
Number analyzed (Participants) | 163
micrograms
  Day 8, ED50, n=157 | 37.4 [17.8 to 57.0]
  Pooled Day 7 and Day 8, ED50, n=160 | 38.2 [14.7 to 61.7]

5. Primary Outcome: Final Dose-response Model Parameter β-FEV1MB-S0 for Trough FEV1
Description: The trough FEV1 data for both the once-daily (QD) and twice-daily (BID) UMEC doses were included in a parametric analysis in order to evaluate dose response. Both a Day 8 dataset and a pooled dataset for Day 7 and Day 8 were analyzed and reported. The rationale for pooling Day 7 and Day 8 (post-hoc analysis) was to ensure informative interpretation of FEV1 response as a function of dose given the repeated measures for trough FEV1 response within each participant on different days. β-FEV1MB-S0 is defined as the covariate (Baseline trough FEV1) effect on the mean Baseline trough FEV1 estimate (S0). FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second.
Time Frame: Day 7 and Day 8 of each treatment period (up to Study Day 50)
Population: as for outcome 1
Measure: Number; unit: fraction of mean estimated Baseline FEV1
Arm/Group | All Study Treatments
Number analyzed (Participants) | 163
fraction of mean estimated Baseline FEV1
  Day 8, βFEV1MB-S0, n=157 | 0.691
  Pooled Day 7 and 8, βFEV1MB-S0, n=160 | 0.686
Statistical Analysis 1: Comparison: All Study Treatments; Test type: Superiority or Other; p < 0.0001, Wald Test — Day 8 analysis
Statistical Analysis 2: Comparison: All Study Treatments; Test type: Superiority or Other; p < 0.0001, Wald Test — Pooled Day 7 and 8 analysis

6. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in One Second (FEV1) on Day 8 of Each Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 on Treatment Day 8 is defined as the value obtained 24 hours after the morning dose administered on Day 7. Analysis was performed using a mixed model with covariates of mean Baseline, period Baseline, treatment, and period as fixed effects and participant as a random effect. Baseline is the FEV1 value recorded pre-dose on Day 1 of each treatment period, mean Baseline is the mean of the Baselines for each participant, and period Baseline is the difference between the Baseline and the mean Baseline in each treatment period for each particiapant. Change from Baseline for each treatment period is the trough FEV1 at Day 8 minus the Baseline value for that treatment period.
Time Frame: Baseline and Day 8 of each treatment period (up to Study Day 50)
Population: mITT Population. All participants with >=1 post-baseline assessment and non-missing covariate data are included in the analysis. The number of participants represents participants who provided data at Day 8.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID | TIO 18 µg QD
Number analyzed (Participants) | 59 | 58 | 56 | 59 | 59 | 55 | 57 | 56
Liters | -0.074 (0.022) | 0.038 (0.022) | 0.027 (0.023) | 0.049 (0.022) | 0.109 (0.022) | 0.051 (0.023) | 0.065 (0.023) | 0.027 (0.023)
Statistical Analysis 1: Comparison: Placebo vs UMEC 15.6 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.113, 95% CI 2-sided [0.058 to 0.168]
Statistical Analysis 2: Comparison: Placebo vs UMEC 31.25 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.101, 95% CI 2-sided [0.045 to 0.158]
Statistical Analysis 3: Comparison: Placebo vs UMEC 62.5 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.124, 95% CI 2-sided [0.068 to 0.179]
Statistical Analysis 4: Comparison: Placebo vs UMEC 125 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.183, 95% CI 2-sided [0.127 to 0.239]
Statistical Analysis 5: Comparison: Placebo vs UMEC 15.6 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.125, 95% CI 2-sided [0.069 to 0.182]
Statistical Analysis 6: Comparison: Placebo vs UMEC 31.25 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.139, 95% CI 2-sided [0.083 to 0.196]
Statistical Analysis 7: Comparison: Placebo vs TIO 18 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.101, 95% CI 2-sided [0.045 to 0.157]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs), defined as those events occuring while participants were on treatment up until one day after the last dose (up to 7 weeks), are reported.
Description: On-treatment SAEs and non-serious AEs were reported for members of the mITT Population, comprised of all participants who were randomized to treatment who had received at least one dose of study medication.
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID | TIO 18 µg QD
Serious Adverse Events (participants affected / at risk) | 0/60 | 1/60 | 1/57 | 0/59 | 0/60 | 0/56 | 0/58 | 0/56
Other Adverse Events (participants affected / at risk) | 2/60 | 3/60 | 0/57 | 0/59 | 8/60 | 4/56 | 1/58 | 2/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=60) | UMEC 15.6 µg QD (N=60) | UMEC 31.25 µg QD (N=57) | UMEC 62.5 µg QD (N=59) | UMEC 125 µg QD (N=60) | UMEC 15.6 µg BID (N=56) | UMEC 31.25 µg BID (N=58) | TIO 18 µg QD (N=56)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=60) | UMEC 15.6 µg QD (N=60) | UMEC 31.25 µg QD (N=57) | UMEC 62.5 µg QD (N=59) | UMEC 125 µg QD (N=60) | UMEC 15.6 µg BID (N=56) | UMEC 31.25 µg BID (N=58) | TIO 18 µg QD (N=56)
Headache (Nervous system disorders) | 2 | 1 | 0 | 0 | 3 | 4 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.